CLINICAL TRIAL: NCT07287215
Title: Investigation of the Relationship Between Motor Imagery Ability and Functional Mobility, Walking, and Balance in Children With Diplegic Cerebral Palsy
Brief Title: Motor Imagery and Functional Performance in Diplegic Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Dilan Demirtaş Karaoba, assistant professor, Inonu University
Other Study IDs: 2025/0725
Record Dates: First submitted 2025-12-02; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Diplegic Cerebral Palsy With Spasticity; Motor İmagery Ability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Motor Imagery Ability Assessment — Laterality Task (Choice Task): Implicit Motor Imagery capacity will be measured through a laterality task, which involves deciding which side a limb belongs to. Right-left discrimination of the foot will be assessed using the "Recognize Foot" application developed by the Neuro Orthopaedic Institute
Other: Mental Stopwatch Paradigm — A mental stopwatch will be used to assess explicit MI capacity. This paradigm compares the time between the actual movement duration and the duration of a similar imagined task.
Other: Functional Mobility — Functional Mobility: Functional Mobility will be assessed using the Functional Mobility Scale (FMS) and the Timed Up and Go test.
Other: Gait assessment: — Gait assessment: The Gillette FDA is a self- or observer-based assessment tool.

SUMMARY:
The main purpose of this study was to examine the relationship between motor imagery capacity and functional mobility, walking and balance in children with diplegic type cerebral palsy.

DETAILED DESCRIPTION:
This study will be conducted using a cross-sectional and correlational screening model to examine the relationship between motor imagery ability and functional mobility, walking, and balance in children with diplegic cerebral palsy. Data collection will be conducted through one-on-one assessments after obtaining written consent from volunteer participants and their families. The data collection tools used in the study are listed below: Demographic Information Form, Motor Imagery Ability Assessment, Mental Stopwatch Paradigm, Functional Mobility, and Gait Assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diplegic CP by a neurologist or pediatric neurologist
* Being between 5 and 18 years of age
* Being between levels I and III on the GMFCS
* Having the cognitive ability to follow the assessment instructions
* Informed consent form has been obtained from the child's family
* The child has agreed to participate voluntarily in the study

Exclusion Criteria:

* Having severe impairments in basic sensory systems such as vision or hearing
* Having additional diagnoses such as epilepsy or autism spectrum disorder
* Demonstrating cognitive or behavioral problems that prevent them from following instructions during the assessment
* Having informed consent from the child's family or the child

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: diplegic cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Mental Stopwatch Paradigm | 24-48 hours
  A mental stopwatch will be used to assess explicit MI capacity. This paradigm compares the time between the actual movement duration and the duration of a similar imagined task.
Laterality Task (Choice Task): | 24-48 hours
  Laterality Task (Choice Task): Implicit Motor Imagery capacity will be measured through a laterality task, which involves deciding which side a limb belongs to. Right-left discrimination of the foot will be assessed using the "Recognize Foot" application developed by the Neuro Orthopaedic Institute
Functional Mobility using the Functional Mobility Scale (FMS) | 24-48 hours
  Functional Mobility: Functional Mobility will be assessed using the Functional Mobility Scale (FMS)
Functional Mobility using the Timed Up and Go test | 24-48 hours
  Functional Mobility: Functional Mobility will be assessed using the Timed Up and Go test.
The Gillette Functional Assessment Questionnaire | 24-48 hours
  Gait assessment: The Gillette Functional Assessment Questionnaire is a self- or observer-based assessment tool, minimum score 22 maximum score 88

CONTACTS AND LOCATIONS:
Locations (1):
- Bingöl, Bingöl, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No